CLINICAL TRIAL: NCT02991118
Title: A Long-term, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy of Bempedoic Acid (ETC-1002) in Patients With Hyperlipidemia at High Cardiovascular Risk Not Adequately Controlled by Their Lipid-Modifying Therapy
Brief Title: Evaluation of Long-Term Efficacy of Bempedoic Acid (ETC-1002) in Patients With Hyperlipidemia at High Cardiovascular Risk
Acronym: CLEAR Wisdom
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-047; 2016-003486-26 (EudraCT Number)
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia; Atherosclerotic Cardiovascular Disease
Keywords: hyperlipidemia; cholesterol; familial hypercholesterolemia; atherosclerotic cardiovascular disease; ASCVD; HeFH; LDL
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis; Hyperlipidemias; Hyperlipoproteinemia Type II | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bempedoic acid (Experimental): bempedoic acid 180 mg/day
  Interventions: Drug: bempedoic acid
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bempedoic acid — bempedoic acid 180 mg tablet taken orally, once daily. Patients remain on ongoing lipid-modifying therapy (not study provided)
  Other Names: ETC-1002
  Arms: bempedoic acid
Drug: placebo — Matching placebo tablet taken orally, once daily. Patients remain on ongoing lipid-modifying therapy (not study provided)
  Other Names: placebo control
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if bemedoic acid (ETC-1002) is effective versus placebo in patients with high cardiovascular risk and elevated LDL cholesterol not adequately controlled by their current therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C ≥100 mg/dL
* High cardiovascular risk (diagnosis of HeFH and/or ASCVD)
* Be on maximally tolerated lipid-modifying therapy (LMT), including maximally tolerated statin either alone or in combination with other LMTs

Exclusion Criteria:

* Total fasting triglyceride ≥500 mg/dL
* Renal dysfunction or nephrotic syndrome or history of nephritis
* Body Mass Index (BMI) ≥50kg/m2
* Significant cardiovascular disease or cardiovascular event in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (2):
- United States (2):
  - Clearwater, Florida
  - Georgetown, Texas

REFERENCES:
- [Background] Goldberg AC, Leiter LA, Stroes ESG, Baum SJ, Hanselman JC, Bloedon LT, Lalwani ND, Patel PM, Zhao X, Duell PB. Effect of Bempedoic Acid vs Placebo Added to Maximally Tolerated Statins on Low-Density Lipoprotein Cholesterol in Patients at High Risk for Cardiovascular Disease: The CLEAR Wisdom Randomized Clinical Trial. JAMA. 2019 Nov 12;322(18):1780-1788. doi: 10.1001/jama.2019.16585. PMID 31714986
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Background] Robinson JG. Management of familial hypercholesterolemia: a review of the recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Manag Care Pharm. 2013 Mar;19(2):139-49. doi: 10.18553/jmcp.2013.19.2.139. PMID 23461430
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Derived] Ballantyne CM, Bays HE, Louie MJ, Smart J, Zhang Y, Ray KK. Factors Associated With Enhanced Low-Density Lipoprotein Cholesterol Lowering With Bempedoic Acid. J Am Heart Assoc. 2022 Aug 2;11(15):e024531. doi: 10.1161/JAHA.121.024531. Epub 2022 Aug 2. PMID 35916348
- [Derived] Banach M, Duell PB, Gotto AM Jr, Laufs U, Leiter LA, Mancini GBJ, Ray KK, Flaim J, Ye Z, Catapano AL. Association of Bempedoic Acid Administration With Atherogenic Lipid Levels in Phase 3 Randomized Clinical Trials of Patients With Hypercholesterolemia. JAMA Cardiol. 2020 Oct 1;5(10):1124-1135. doi: 10.1001/jamacardio.2020.2314. PMID 32609313
- See also: World Health Organization Fact Sheet No. 317 — http://www.who.int/mediacentre/factsheets/fs317/en/
- See also: What Is Familial Hypercholesterolemia — https://thefhfoundation.org/about-fh/what-is-fh/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 779 participants were randomized 2:1 to receive either bempedoic acid or placebo.
Pre-assignment Details: The study consisted of 3 periods: a 1-week screening period; a 4-week single-blind, placebo run-in period; and a 52-week double-blind, randomized treatment period.
Groups:
- Placebo: Participants received a placebo tablet once daily by mouth for 4 weeks prior to the 52-week double-blind treatment period. During the treatment period, participants received placebo once daily by mouth for 52 weeks. Participants remained on ongoing lipid-modifying therapy (not study provided) throughout the study.
- Bempedoic Acid: Participants received a placebo tablet once daily by mouth for 4 weeks prior to the 52-week double-blind treatment period. During the treatment period, participants received a bempedoic acid 180 milligram (mg) tablet once daily by mouth for 52 weeks. Participants remained on ongoing lipid-modifying therapy (not study provided) throughout the study.
Period: Overall Study
Arm/Group | Placebo | Bempedoic Acid
Started | 257 | 522
Completed | 250 | 490
Not Completed | 7 | 32
Not completed — Death | 3 | 8
Not completed — Protocol Violation | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Moved out of the country | 0 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Could not attend study visits | 0 | 1
Not completed — Lost to Follow-up | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bempedoic Acid | Total
Number analyzed (Participants) | 257 | 522 | 779
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.73) | 64.1 (8.82) | 64.3 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 194 | 283
  Male | 168 | 328 | 496
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 4 | 4
  Black or African American | 12 | 24 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 244 | 491 | 735
  Multiple | 0 | 2 | 2
Mean low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1.
  milligrams per deciliter (mg/dL) | 122.4 (38.30) | 119.4 (37.75) | 120.43 (37.931)
LDL-C category [Count of Participants; unit: Participants]
  <130 mg/dL | 173 | 365 | 538
  ≥130 and <160 mg/dL | 45 | 89 | 134
  ≥160 mg/dL | 39 | 68 | 107
Mean non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the non-HDL-C values from the last two non-missing values on or prior to Day 1.
  mg/dL | 153.7 (44.36) | 150.7 (42.75) | 151.7 (43.28)
Mean total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the TC values from the last two non-missing values on or prior to Day 1.
  mg/dL | 204.8 (46.06) | 202.1 (42.71) | 203.0 (43.83)
Mean apolipoprotein B (apoB) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing value on or prior to Day 1.
  mg/dL | 118.6 (30.53) | 116.2 (29.58) | 117.0 (29.90)
Median high-sensitivity C-reactive protein (hsCRP) [Median (Inter-Quartile Range); unit: milligrams per Liter] — Baseline was defined as the last non-missing value on or prior to Day 1. Dispersion data are reported as the first quartile and third quartile values.
  milligrams per Liter | 1.880 [0.920 to 3.790] | 1.610 [0.870 to 3.455] | 1.700 [0.870 to 3.560]
Median triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 143.00 [106.00 to 189.00] | 139.25 [102.50 to 190.00] | 140.00 [103.00 to 189.50]
Concomitant lipid-modifying therapy (LMT) medications [Count of Participants; unit: Participants] — Concomitant medications were defined as medications that were ongoing at the time of double-blind investigational medicinal product (IMP) initiation or new medications that started after double-blind IMP initiation and within 30 days following the date of the last dose of IMP. Other LMT included ezetimibe, fish oil, omega-3 fatty acids, omega-3-acid ethyl ester, alirocumab, evolocumab, and kolestop. Data are reported for participants who took at least one concomitant LMT.
  Participants
    Statins | 232 | 478 | 710
    Fibrates | 17 | 26 | 43
    Nicotinic acid and derivatives | 0 | 1 | 1
    Other lipidmodifying therapies | 38 | 63 | 101
    Bile acid sequestrants | 3 | 5 | 8
History of atherosclerotic cardiovascular disease (ASCVD) [Count of Participants; unit: Participants] — Data for participants with ASCVD only (without heterozygous familial hypercholesterolemia [HeFH]) are reported.
  Participants | 241 | 495 | 736
History of HeFH [Count of Participants; unit: Participants] — Data for participants with HeFH (with or without ASCVD) are reported.
  Participants | 16 | 27 | 43
History of impaired fasting glucose [Count of Participants; unit: Participants] | 5 | 9 | 14
Background LMT [Count of Participants; unit: Participants]
  Statins with or without other LMTs | 228 | 470 | 698
  Statins without other LMTs | 196 | 416 | 612
  Statins with other LMTs | 32 | 54 | 86
  Other LMTs without statins | 15 | 22 | 37
  No LMT or statin | 14 | 30 | 44
Disease history [Count of Participants; unit: Participants] — The presence of these conditions was determined by participant-reported medical history.
  Participants
    Hypertension | 224 | 438 | 662
    Coronary heart disease | 205 | 432 | 637
    Diabetes | 81 | 155 | 236
    Impaired fasting glucose | 5 | 9 | 14
Body mass index (BMI) [Mean (Standard Deviation); unit: kilograms per meters squared (kg/m^2)] — BMI was calculated as weight in kilograms divided by height in meters squared.
  kilograms per meters squared (kg/m^2) | 30.64 (5.048) | 30.01 (5.192) | 30.22 (5.150)
Estimated glomerular filtration rate (eGFR) category [Count of Participants; unit: Participants] — eGFR was measured in milliliters per minutes per 1.73 meters squared (mL/min/1.73 m^2).
  Participants
    ≥90 mL/min/1.73 m^2 | 56 | 107 | 163
    ≥60 to <90 mL/min/1.73 m^2 | 164 | 338 | 502
    <60 mL/min/1.73 m^2 | 37 | 77 | 114
Statin intensity [Count of Participants; unit: Participants] — Baseline statin intensity were based on stratification at randomization. Low-intensity statins: simvastatin 10 milligrams (mg); pravastatin 10-20 mg; lovastatin 20 mg; fluvastatin 20-40 mg; pitavastatin 1 mg. Moderate-intensity statins: atorvastatin 10-20 mg; rosuvastatin 5-10 mg; simvastatin 20 mg; pravastatin 40-80 mg; lovastatin 40 mg; fluvastatin XL 80 mg; fluvastatin 40 mg twice a day; pitavastatin 2-4 mg. High-intensity statins: atorvastatin 40-80 mg; rosuvastatin 20-40 mg.
  Participants
    Low intensity or no statin | 40 | 78 | 118
    Moderate intensity | 82 | 166 | 248
    High intensity | 135 | 278 | 413
Numer of participants receiving ezetimibe [Count of Participants; unit: Participants] | 24 | 39 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Baseline is defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in LDL-C was analyzed using an analysis of covariance (ANCOVA) model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (atherosclerotic cardiovascular diseases [ASCVD] and heterozygous familial hypercholesterolemia [HeFH]) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate. In the ANCOVA model, missing LDL-C data at Week 12 are imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Baseline; Week 12
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 257 | 522
percent change | 2.35 (1.446) | -15.07 (1.073)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -17.42, 95% CI 2-sided [-20.951 to -13.896], Standard Error of Mean 1.800

2. Secondary Outcome: Percent Change From Baseline to Week 24 in LDL-C
Description: Baseline is defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in LDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate. In the ANCOVA model, missing LDL-C data at Week 24 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Baseline; Week 24
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 257 | 522
percent change | 2.66 (1.910) | -12.10 (1.479)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -14.77, 95% CI 2-sided [-19.504 to -10.027], Standard Error of Mean 2.418

3. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Baseline is defined as the mean of the non-HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in non-HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate. In the ANCOVA model, missing non-HDL-C data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Baseline; Week 12
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 257 | 522
percent change | 2.28 (1.351) | -10.75 (0.952)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -13.03, 95% CI 2-sided [-16.270 to -9.794], Standard Error of Mean 1.652

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol (TC)
Description: Baseline is defined as the mean of the TC values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in TC was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate. In the ANCOVA model, missing TC data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Baseline; Week 12
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 257 | 522
percent change | 1.26 (1.010) | -9.94 (0.688)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -11.20, 95% CI 2-sided [-13.599 to -8.801], Standard Error of Mean 1.224

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein b (Apo B)
Description: Baseline for apo B was defined as the last non-missing value on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in apo B was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate. In the ANCOVA model, missing apo B data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Baseline; Week 12
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 257 | 522
percent change | 3.73 (1.340) | -9.29 (0.851)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -13.02, 95% CI 2-sided [-16.130 to -9.907], Standard Error of Mean 1.587

6. Secondary Outcome: Percent Change From Baseline to Week 12 in High-sensitivity C-reactive Protein (hsCRP)
Description: Baseline for hsCRP was defined as the last non-missing value on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 240 | 467
percent change | -9.366 [-36.320 to 35.241] | -18.699 [-46.067 to 23.864]
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.039, Wilcoxon Rank Sum Test; Location shift = -8.733, 95% CI 2-sided [-17.238 to -0.434] — The location shift and asymptotic 95% confidence interval are based on Hodges-Lehman estimation

7. Secondary Outcome: Change From Baseline to Week 12 in LDL-C
Description: Baseline is defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Change from Baseline is calculated as the post-baseline value minus the baseline value. Analysis was conducted using descriptive statistics by treatment group using observed data.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 253 | 498
mg/dL | 0.0 (30.62) | -21.2 (30.82)

8. Secondary Outcome: Change From Baseline to Week 24 in LDL-C
Description: as for outcome 7
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 247 | 485
mg/dL | -1.0 (37.51) | -18.7 (35.76)

9. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in Triglycerides (TGs)
Description: Baseline is defined as the mean of the TG values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in TG was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 253 | 499
percent change | 6.12 (2.294) | 11.01 (2.312)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p = 0.134, ANCOVA; Difference in LS mean = 4.89, 95% CI 2-sided [-1.504 to 11.292], Standard Error of Mean 3.258

10. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in HDL-C
Description: Baseline is defined as the mean of the HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 253 | 499
percent change | -0.25 (0.864) | -6.38 (0.741)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -6.13, 95% CI 2-sided [-8.369 to -3.896], Standard Error of Mean 1.139

11. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in LDL-C
Description: Baseline was defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in LDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 237 | 467
percent change | -0.97 (1.830) | -13.24 (1.412)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -12.27, 95% CI 2-sided [-16.813 to -7.722], Standard Error of Mean 2.314

12. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in Non-HDL-C
Description: Baseline was defined as the mean of the non-HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in non-HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate.
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 247 | 485
percent change | 2.44 (1.611) | -10.19 (1.200)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -12.63, 95% CI 2-sided [-16.580 to -8.682], Standard Error of Mean 2.010

13. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in Non-HDL-C
Description: as for outcome 12
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 237 | 467
percent change | -0.42 (1.605) | -10.34 (1.150)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -9.92, 95% CI 2-sided [-13.803 to -6.037], Standard Error of Mean 1.976

14. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in TC
Description: Baseline was defined as the mean of the TC values from the last two non-missing values on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in TC was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate.
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 247 | 486
percent change | 1.52 (1.216) | -9.25 (0.857)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -10.77, 95% CI 2-sided [-13.698 to -7.848], Standard Error of Mean 1.489

15. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in TC
Description: as for outcome 14
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 237 | 467
percent change | -1.89 (1.199) | -10.25 (0.828)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -8.36, 95% CI 2-sided [-11.223 to -5.493], Standard Error of Mean 1.458

16. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in Apo B
Description: Baseline for apo B was defined as the last non-missing value on or prior to Day 1. Percent change from Baseline is calculated as ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. Percent change from Baseline in apo B was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and Baseline as a covariate.
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 144 | 294
percent change | 4.39 (2.090) | -8.61 (1.267)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -13.00, 95% CI 2-sided [-17.829 to -8.175], Standard Error of Mean 2.451

17. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in Apo B
Description: as for outcome 16
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 237 | 464
percent change | 3.01 (1.502) | -6.56 (0.983)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -9.58, 95% CI 2-sided [-13.107 to -6.047], Standard Error of Mean 1.796

18. Other Pre Specified Outcome: Percent Change From Baseline to Week 24 in hsCRP
Description: as for outcome 6
Time Frame: Baseline; Week 24
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 127 | 271
percent change | 1.563 [-32.174 to 47.500] | -24.107 [-51.502 to 14.035]
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, Wilcoxon Rank Sum Test; Location shift = -21.278, 95% CI 2-sided [-32.250 to -10.034] — The location shift and asymptotic 95% confidence interval are based on Hodges-Lehman estimation

19. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in hsCRP
Description: as for outcome 6
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 237 | 465
percent change | -6.250 [-39.286 to 41.810] | -16.727 [-50.877 to 31.429]
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p = 0.102, Wilcoxon Rank Sum Test; Location shift = -7.587, 95% CI 2-sided [-16.978 to 1.653] — The location shift and asymptotic 95% confidence interval are based on Hodges-Lehman estimation

20. Other Pre Specified Outcome: Change From Baseline to Week 52 in LDL-C
Description: Baseline was defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Change from Baseline is calculated as the post-baseline value minus the baseline value. Analysis was conducted using descriptive statistics by treatment group using observed data. Change from Baseline in LDL-C was analyzed using an ANCOVA model with change from baseline as the dependent variable, treatment, cardiovascular risk (ASCVD and HeFH) crossed with Baseline statin intensity (low/moderate and high) as fixed effects and baseline as a covariate.
Time Frame: Baseline; Week 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 237 | 467
mg/dL | -4.71 (2.216) | -19.78 (1.433)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -15.07, 95% CI 2-sided [-20.260 to -9.878], Standard Error of Mean 2.641

ADVERSE EVENTS:
Time Frame: up to Week 52
Description: Treatment-emergent events, defined as those adverse events that began or worsened after the first dose of investigational medicinal product (IMP) until 30 days after the last dose of IMP, were collected and reported. The analysis was performed using the Safety Analysis Set, comprised of all randomized participants who received >=1 dose of IMP.
Groups:
- Placebo: Participants received placebo tablet once daily by mouth for 4 weeks prior to the 52-week double-blind treatment period. During the treatment period, participants received placebo once daily by mouth for 52 weeks. Participants remained on ongoing lipid-modifying therapy (not study provided) throughout the study.
Arm/Group | Placebo | Bempedoic Acid
All-Cause Mortality (participants affected / at risk) | 2/257 | 6/522
Serious Adverse Events (participants affected / at risk) | 48/257 | 106/522
Other Adverse Events (participants affected / at risk) | 88/257 | 211/522
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=257) | Bempedoic Acid (N=522)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 1 | 12
Angina unstable (Cardiac disorders) | 6 | 9
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 4
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 4
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 6 | 7
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 4 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
Exercise tolerance decreased (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urethral stricture post infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Gas poisoning (Injury, poisoning and procedural complications) | 0 | 1
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 3
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 4
Post stroke epilepsy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 4
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Perinephritis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Supportive care (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Subclavian artery thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=257) | Bempedoic Acid (N=522)
Anaemia (Blood and lymphatic system disorders) | 3 | 14
Diarrhoea (Gastrointestinal disorders) | 7 | 16
Fatigue (General disorders) | 9 | 6
Bronchitis (Infections and infestations) | 6 | 7
Lower respiratory tract infection (Infections and infestations) | 7 | 7
Nasopharyngitis (Infections and infestations) | 13 | 27
Upper respiratory tract infection (Infections and infestations) | 9 | 19
Urinary tract infection (Infections and infestations) | 5 | 24
Blood uric acid increased (Investigations) | 1 | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 10
Gout (Metabolism and nutrition disorders) | 2 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 22
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 7 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 15
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 11
Dizziness (Nervous system disorders) | 9 | 8
Headache (Nervous system disorders) | 7 | 10
Hypertension (Vascular disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02991118/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02991118/SAP_001.pdf